CLINICAL TRIAL: NCT05252351
Title: Cardiac Imaging in Congenital Aortic Stenosis - Unravelling Risk Factors and Predicting Clinical Outcome
Brief Title: Cardiac Imaging in Adults With Congenital Aortic Stenosis
Acronym: CAS
Status: Active, not recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Principal Investigator, Dr. Annemien E. van den Bosch, Principal Investigator, Erasmus Medical Center
Other Study IDs: CAS study
Record Dates: First submitted 2022-01-17; First posted 2022-02-23 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Congenital Aortic Stenosis
Keywords: Congenital Aortic Stenosis; Bicuspid Aortic Valve; Left ventricular function; Cardiac imaging; Myocardial tissue characterization
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with congenital aortic stenosis

SUMMARY:
The CAS study is a prospective observational cohort study investigating the effects of congenital aortic stenosis (ConAoS) on the left ventricular function and the prevalence, pattern and expanse of left ventricular hypertrophy (LVH), myocardial stiffness and myocardial fibrosis.

DETAILED DESCRIPTION:
Congenital aortic stenosis (ConAoS) accounts for 4-8% of all congenital cardiac diagnoses. It is often caused by a bicuspid aortic valve (BAV), which has an estimated prevalence of 0.5-2% in the general population. Patients with ConAoS may remain asymptomatic, but gradual deterioration of the stenosis and the strong association of BAV with aortic dilatation contributes to important morbidity and mortality. The prevalent nature of this heart defect implies an important health problem resulting in hospitalization and (re-) interventions. As it is still largely unknown which markers predict adverse outcome, the aim of this study is to evaluate trends in imaging and biomarkers in this patient population and their relation with clinical outcome.

It is increasingly acknowledged that aortic stenosis is not only a disease of the valve, but also of the left ventricle (LV) and the aorta. In the course of disease progression, pressure overload and ventricular wall stress lead to remodeling of the LV, which eventually leads to left ventricular hypertrophy (LVH) and myocardial fibrosis. Although these processes have been described in patients with aortic stenosis, little is known about the prevalence and prognostic relevance of LVH and myocardial fibrosis in patients with ConAoS, who are often relatively young. Applying upcoming innovative imaging modalities such as high frame rate echocardiography and T1-mapping in patients with ConAoS will increase our knowledge on tissue characterization, which in turn will facilitate identifying patients at high risk for complications and rapid disease progression.

The CAS study is a clinical observational study investigating the effects of ConAoS on the left ventricular function and the prevalence, pattern and expanse of LVH, myocardial stiffness and myocardial fibrosis. Moreover, the prognostic capacity of the presence of these pathological processes will be assessed, correlating findings at baseline to clinical outcome by assessing the occurrence of cardiovascular events and all-cause mortality during 3-year clinical follow-up. The investigators will unravel biomarker and imaging predictors for myocardial dysfunction (systolic and diastolic) with specific attention for male-female differences. This newly gained knowledge will enable the investigators to improve and individualize current treatment protocols and derive novel therapeutic strategies for adult patients with ConAoS.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet the following criteria:

* Aged ≥ 18 years
* Capable of understanding and signing informed consent.

Inclusion criteria for the CAS study are patients diagnosed with a valvular congenital aortic stenosis. Two groups of patients will be included:

* Patients with a prior aortic valve replacement (AVR)
* Patients without a prior AVR and with an aortic jet velocity ≥ 2.5 m/s.

Exclusion Criteria:

* Patients with severe aortic regurgitation
* Presence of any of the following contra-indications for MRI

  * Contra-indication to gadolinium based contrast media (eGFR <30 ml/min or contrast allergy)
  * Other contra-indications such as presence of pacemaker/implantable cardioverter defibrillator, severe claustrophobia or pregnancy
* Patients known with or previously treated because of aortic coarctation.
* Patients known with genetic syndromes or connective tissue disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult ConAoS patients, who are visiting the outpatient clinic of the Erasmus MC.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of myocardial fibrosis | Baseline
  Assessed at baseline using cardiovascular magnetic resonance imaging (late gadolinium enhancement (LGE) and T1 mapping pre- and post-contrast)

SECONDARY OUTCOMES:
Left ventricular function | Baseline
  This outcome is measured by strain measurements using echocardiography and cardiovascular magnetic resonance imaging (CMR)
Shear wave velocity | Baseline
  Shear wave velocity is measured using high frame rate echocardiography
Physical activity in daily life | Baseline
  This outcome is measured by the following questionnaire: Short Questionnaire to Assess Health-enhancing physical activity (SQUASH)
Quality of life (SF-36) | Baseline
  This outcome is assessed by using the SF-36 questionnaire
Occurence of ventricular arrhythmias | Baseline
  This outcome is assessed by the occurence of ventricular ectopies and non-sustained ventricular tachycardia (VT) on Holter ECG for 48 hours.
Conduction abnormalities on ECG | Baseline
  For this outcome the conduction times on ECG will be measured
All-cause mortality | 3 years
Cardiovascular events | 3 years
  Incidents of heart failure, arrhythmias, endocarditis, aortopathy (aortic dissection and/or aortic aneurysm), (re-) interventions and (re-) operations of the aortic valve and/or ascending aorta and hospitalizations for other cardiac reasons
Aortic flow patterns | Baseline
  This outcome is measured using 4D flow CMR
Blood biomarkers | Baseline
Fear of movement | Baseline
  This outcome is measured using the following questionnaire: Tampa Scale for Kinesiophobia (TSK-NL Heart)

CONTACTS AND LOCATIONS:
Overall Officials: Annemien E van den Bosch, MD, PHD, Principal Investigator — Erasmus Medical Center; Alexander Hirsch, MD, PHD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands